CLINICAL TRIAL: NCT03829319
Title: A Phase 3 Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of Pemetrexed + Platinum Chemotherapy + Pembrolizumab (MK-3475) With or Without Lenvatinib (E7080/MK-7902) as First-line Intervention in Participants With Metastatic Nonsquamous Non-small Cell Lung Cancer (LEAP-006)
Brief Title: Safety and Efficacy Study of Pemetrexed + Platinum Chemotherapy + Pembrolizumab (MK-3475) With or Without Lenvatinib (MK-7902/E7080) as First-line Intervention in Adults With Metastatic Nonsquamous Non-small Cell Lung Cancer (MK-7902-006/E7080-G000-315/LEAP-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7902-006; MK-7902-006 (Other: MSD Protocol Number); E7080-G000-315 (Other: Eisai Protocol Number); LEAP-006 (Other: MSD); 194658 (Registry Identifier: JAPIC-CTI); 2018-003824-35 (EudraCT Number)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Nonsquamous Non-small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Cisplatin; Pemetrexed; lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib (Experimental): Participants receive carboplatin Area Under Curve 5 mg/mL/min (AUC5) or cisplatin 75 mg/m^2 via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS lenvatinib via oral capsule once daily.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Lenvatinib
- Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo (Placebo Comparator): In Parts 1 and 2: Participants receive carboplatin AUC5 or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS (Part 2 only) placebo matching lenvatinib via oral capsule once daily.
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Placebo matching lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion Q3W
  Other Names: MK-3475
Drug: Carboplatin — IV infusion Q3W
Drug: Cisplatin — IV infusion Q3W
Drug: Pemetrexed — IV infusion Q3W
Drug: Lenvatinib — Oral capsule once daily
  Other Names: MK-7902; E7080
  Arms: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Lenvatinib
Drug: Placebo matching lenvatinib — Oral capsule once daily
  Arms: Pemetrexed+Platinum Chemotherapy+Pembrolizumab+Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pemetrexed + platinum chemotherapy + pembrolizumab (MK-3475) with or without lenvatinib (MK-7902/E7080) as first-line intervention in adults with metastatic nonsquamous non-small cell lung cancer.

The primary study hypotheses state that: 1) the combination of lenvatinib + platinum doublet chemotherapy + pembrolizumab prolongs Progression-free Survival (PFS) as assessed by blinded independent central review (BICR) per modified Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST 1.1) compared to matching placebo + platinum doublet chemotherapy + pembrolizumab, and 2) the combination of lenvatinib + platinum doublet chemotherapy + pembrolizumab prolongs Overall Survival (OS) compared to matching placebo + platinum doublet chemotherapy + pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IV (American Joint Committee on Cancer [AJCC], version 8 or current version), nonsquamous NSCLC.
* Confirmation that Epidermal Growth Factor Receptor (EGFR), ALK Receptor Tyrosine Kinase (ALK), or ROS1 Receptor Tyrosine Kinase (ROS1)-directed therapy is not indicated as primary treatment (documentation of absence of tumor-activating EGFR mutations AND absence of ALK and ROS1 gene rearrangements OR presence of a Kirsten Rat Sarcoma (KRAS) gene mutation).
* Have measurable disease based on RECIST 1.1. Note: Lesions that appear measurable, but are situated in a previously irradiated area, can be considered measurable (eligible for selection as target lesions) if they have shown documented growth since the completion of radiation.
* Provided an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion (not previously irradiated).
* Life expectancy of at least 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days prior to the first dose of study intervention but before randomization.
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions is more stringent than the requirements above, the local label requirements are to be followed.
* Male participants must agree for at least 7 days after the last dose of lenvatinib/matching placebo and up to 180 days after the last dose of chemotherapeutic agents to:

  1. Refrain from donating sperm PLUS either:
  2. Be abstinence from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR
  3. Must agree to use contraception unless confirmed to be azoopsermic (vasectomized or secondary to medical cause) as detailed below:

     1. Agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant Note: Men with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile-vaginal penetration.

Note: 7 days after lenvatinib/matching placebo is stopped, if the participant is on pembrolizumab only and is greater than 180 days post chemotherapy, no male contraception measures are needed.

* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  1. Is not a WOCBP OR
  2. Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 120 days post pembrolizumab and/or 30 days post-lenvatinib/matching placebo, and up to 180 days post last dose of chemotherapeutic agents, whichever occurs last.
* Adequate organ function.
* Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week prior to randomization. Note: Participants must not have a history of uncontrolled or poorly-controlled hypertension, defined as >150/90 mm Hg for >4 weeks despite standard medical management.

Exclusion Criteria:

* Known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, clinically stable, and have not required steroids for at least 14 days prior to the first dose of study intervention.
* History of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.
* Radiographic evidence of intratumoral caviations, encasement, or invasion of a major blood vessel. Additionally, the degree of proximity to major blood vessels should be considered for exclusion because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis after lenvatinib-therapy. (In the chest, major blood vessels include the main pulmonary artery, the left and right pulmonary arteries, the 4 major pulmonary veins, the superior or inferior vena cava, and the aorta).
* Known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy. Note: The time requirement also does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study intervention.
* Has had allogeneic tissue/solid organ transplant.
* Known history of human immunodeficiency virus (HIV) infection. HIV testing is not required unless mandated by the local health authority.
* Known history of Hepatitis B or active Hepatitis C. No testing for Hepatitis B or Hepatitis C is required unless mandated by the local health authority.
* History of a gastrointestinal condition or procedure that in the opinion of the investigator may affect oral drug absorption.
* Active hemoptysis (at least 0.5 teaspoon of bright red blood) within 2 weeks prior to the first dose of study intervention.
* Significant cardiovascular impairment within 12 months prior to the first dose of study intervention, including history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction, cerebrovascular accident (CVA)/stroke, or cardiac arrhythmia associated with hemodynamic instability.
* Known history of active tuberculosis.
* Active infection requiring systemic therapy.
* Has not recovered adequately from any toxicity and/or complication from major surgery prior to the first dose of study intervention.
* Previously had a severe hypersensitivity reaction to treatment with a monoclonal antibody or has a known sensitivity to any component of lenvatinib or pembrolizumab, or as applicable, carboplatin, cisplatin, or pemetrexed.
* A WOCBP who has a positive urine pregnancy test within 24 hours prior to randomization or treatment allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
* Received prior systemic chemotherapy or other targeted or biological antineoplastic therapy for their metastatic NSCLC. Note: Prior treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic NSCLC.
* Received prior treatment with pembrolizumab or any other anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2 agent, with lenvatinib or any other receptor tyrosine kinase inhibitor (RTKi), or with an agent directed to another stimulatory or co-inhibitory T cell receptor.
* Received radiotherapy within 14 days prior to the first dose of study intervention or received lung radiation therapy of >30 Gy within 6 months prior to the first dose of study intervention. Note: Participants must have recovered from all radiation-related toxicities to Grade ≤1, not required corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Received systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of study intervention.
* Received a live or live attenuated vaccine within 30 days prior to the first dose of study intervention. Note: killed vaccines are allowed.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a prolongation of QTc interval (calculated using Fridericia's formula) of >480 msecl.
* Left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
* Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (158):
- United States (17):
  - El Camino Hospital Cancer Center ( Site 0529), Mountain View, California
  - Yale University ( Site 0519), New Haven, Connecticut
  - Holy Cross Hospital ( Site 0512), Fort Lauderdale, Florida
  - Mercy Health-Paducah Medical Oncology and Hematology ( Site 0570), Paducah, Kentucky
  - Henry Ford Health System ( Site 0563), Detroit, Michigan
  - Saint Lukes Cancer Institute ( Site 0541), Kansas City, Missouri
  - Broome Oncology, LLC ( Site 0562), Johnson City, New York
  - Sanford Health Roger Maris Cancer Center ( Site 0533), Fargo, North Dakota
  - Stephenson Cancer Center ( Site 0504), Oklahoma City, Oklahoma
  - Good Samaritan Hospital Corvallis ( Site 0521), Corvallis, Oregon
  - Thomas Jefferson University Hospital ( Site 0548), Philadelphia, Pennsylvania
  - Abington Hospital - Asplundh Cancer Center ( Site 0575), Willow Grove, Pennsylvania
  - West Cancer Center - East Campus ( Site 0544), Germantown, Tennessee
  - Parkland Health & Hospital System ( Site 0576), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0558), Dallas, Texas
  - Utah Cancer Specialists ( Site 0523), Salt Lake City, Utah
  - West Virginia University ( Site 0526), Morgantown, West Virginia
- Argentina (8):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 0367), Berazategui, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata ( Site 0371), Mar del Plata, Buenos Aires
  - CEMIC ( Site 0370), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 0365), Rosario, Santa Fe Province
  - Hospital Aleman ( Site 0368), Buenos Aires
  - Instituto Medico Especializado Alexander Fleming ( Site 0369), Buenos Aires
  - CEMAIC ( Site 0374), Córdoba
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica ( Site 0372), San Juan
- Australia (7):
  - Blacktown Hospital Western Sydney Local Health District ( Site 0008), Blacktown, New South Wales
  - Port Macquarie Base Hospital ( Site 0001), Port Macquarie, New South Wales
  - Chris OBrien Lifehouse ( Site 0006), Sydney, New South Wales
  - Westmead Hospital ( Site 0009), Sydney, New South Wales
  - Cairns Hospital ( Site 0002), Cairns, Queensland
  - The Prince Charles Hospital ( Site 0010), Chermside, Queensland
  - Ballarat Health Services ( Site 0003), Ballarat, Victoria
- Canada (9):
  - Moncton Hospital - Horizon Health Network ( Site 0410), Moncton, New Brunswick
  - Juravinski Cancer Centre ( Site 0407), Hamilton, Ontario
  - Kingston Health Sciences Centre ( Site 0414), Kingston, Ontario
  - Lakeridge Health ( Site 0406), Oshawa, Ontario
  - Sault Area Hospital ( Site 0413), Sault Ste. Marie, Ontario
  - Hopital Cite de la Sante de Laval ( Site 0400), Laval, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0412), Montreal, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec ( Site 0403), Québec, Quebec
  - CIUSSS de la Mauricie et du Centre du Quebec ( Site 0408), Trois-Rivières, Quebec
- Chile (8):
  - Clinica Universidad Catolica del Maule ( Site 0385), Talca, Maule Region
  - OrlandiOncologia ( Site 0381), Santiago, Region M. de Santiago
  - Fundacion Arturo Lopez Perez FALP ( Site 0383), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0382), Santiago, Region M. de Santiago
  - Bradford Hill Centro de Investigaciones Clinicas ( Site 0387), Santiago, Region M. de Santiago
  - Centro de Investigacion y desarrollo Oncologico SpA - CIDO SpA ( Site 0380), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0384), Viña del Mar, Región de Valparaíso
  - Centro Oncologico Antofagasta ( Site 0386), Antofagasta
- China (19):
  - Peking Union Medical College Hospital ( Site 0108), Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Science ( Site 0117), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0120), Beijing, Beijing Municipality
  - The Second Hospital Affiliated to AMU ( Site 0119), Chongqing, Chongqing Municipality
  - First Affiliated Hospital of The Third Military Medical University ( Site 0118), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0102), Fuzhou, Fujian
  - Southern Medical University Nanfang Hospital ( Site 0121), Guangzhou, Guangdong
  - The Third Affiliated Hospital of Harbin Medical University ( Site 0100), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0112), Zhengzhou, Henan
  - Wuhan Union Hospital Cancer Center-Cancer Center ( Site 0123), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0122), Wuhan, Hubei
  - Jilin Cancer Hospital ( Site 0115), Changchun, Jilin
  - Zhongshan Hospital Fudan University ( Site 0103), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 0101), Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0111), Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 0110), Urumuqi, Xinjiang
  - The First Affiliated Hospital Zhejiang University ( Site 0109), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0113), Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University ( Site 0124), Wenzhou, Zhejiang
- France (9):
  - Hopital Cardiologique Louis Pradel ( Site 0141), Bron, Auvergne-Rhône-Alpes
  - Centre Paul Strauss ( Site 0144), Strasbourg, Bas-Rhin
  - Hopital Nord du Marseille ( Site 0147), Marseille, Bouches-du-Rhone
  - Hopital Foch ( Site 0145), Suresnes, Hauts-de-Seine
  - Centre de Cancerologie du Grand Montpellier ( Site 0142), Montpellier, Herault
  - Hopital Laennec ( Site 0146), Nantes, Loire-Atlantique
  - Hopital Robert Schuman ( Site 0143), Vantoux, Moselle
  - L'hopital Nord-Ouest - Centre Hospitalier de Villefranche sur Saone ( Site 0149), Villefranche-sur-Saône, Rhone
  - Hopital Cochin ( Site 0140), Paris
- Germany (8):
  - Klinikum Esslingen GmbH ( Site 0164), Esslingen am Neckar, Baden-Wurttemberg
  - Krankenhaus Nordwest ( Site 0169), Frankfurt am Main, Hesse
  - Pius Hospital Oldenburg ( Site 0170), Oldenburg, Lower Saxony
  - Uniklinik RWTH Aachen ( Site 0160), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes ( Site 0165), Homburg, Saarland
  - Krankenhaus Martha Maria Halle-Doelau ( Site 0166), Halle, Saxony-Anhalt
  - LungenClinic Grosshansdorf GmbH ( Site 0171), Großhansdorf, Schleswig-Holstein
  - Hamato-Onkologie Hamburg Prof. Laack und Partner ( Site 0161), Hamburg
- Israel (9):
  - Soroka Medical Center ( Site 0222), Beersheba
  - Rambam Medical Center ( Site 0223), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 0229), Jerusalem
  - Meir Medical Center ( Site 0221), Kfar Saba
  - Holy Family Hospital ( Site 0228), Nazareth
  - Rabin Medical Center ( Site 0224), Petah Tikva
  - Sheba Medical Center ( Site 0220), Ramat Gan
  - Sourasky Medical Center ( Site 0225), Tel Aviv
  - Shamir Medical Center-Assaf Harofeh ( Site 0227), Ẕerifin
- Japan (11):
  - National Hospital Organization Nagoya Medical Center ( Site 0017), Nagoya, Aichi-ken
  - Fujita Health University Hospital ( Site 0016), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 0024), Kashiwa, Chiba
  - Kanazawa University Hospital ( Site 0018), Kanazawa, Ishikawa-ken
  - Osaka Habikino Medical Center ( Site 0020), Habikino, Osaka
  - Kansai Medical University Hospital ( Site 0022), Hirakata, Osaka
  - Niigata Cancer Center Hospital ( Site 0019), Niigata
  - National Cancer Center Hospital ( Site 0026), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0015), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0021), Tokyo
  - Wakayama Medical University Hospital ( Site 0025), Wakayama
- New Zealand (2):
  - Tauranga Hospital ( Site 0004), Tauranga, Bay of Plenty
  - Auckland City Hospital ( Site 0011), Auckland
- Poland (6):
  - Pleszewskie Centrum Medyczne w Pleszewie Sp. z o.o. ( Site 0615), Pleszew, Greater Poland Voivodeship
  - MED-POLONIA Sp. z o.o. ( Site 0609), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im.prof. F. Lukaszczyka w Bydgoszczy ( Site 0601), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0603), Warsaw, Masovian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 0602), Koszalin, West Pomeranian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii ( Site 0613), Lodz, Łódź Voivodeship
- Russia (11):
  - Leningrad Regional Oncology Center ( Site 0271), Saint Petersburg, Leningradskaya Oblast'
  - City Clinical Hospital 1 na. NI. Pirogov ( Site 0270), Moscow, Moscow
  - Central Clinical Hospital with outpatient Clinic ( Site 0262), Moscow, Moscow
  - National Medical Research Radiology Centre ( Site 0260), Moscow, Moscow
  - FSAI Treatment and Rehabilitation Centre of the MoH and SD of RF ( Site 0264), Moscow, Moscow
  - Moscow Regional Oncological Dispensary ( Site 0274), Balashikha, Moscow Oblast
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 0272), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 0267), Omsk, Omsk Oblast
  - First Pavlov State Medical University of Saint Petersburg-Department of Oncology ( Site 0273), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0269), Saint Petersburg, Sankt-Peterburg
  - SAHI Republican Clinical Oncological Dispensary of the MoH of RT ( Site 0261), Kazan', Tatarstan, Respublika
- South Korea (4):
  - National Cancer Center ( Site 0061), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 0064), Gyeonggi-do, Kyonggi-do
  - Chungbuk National University Hospital ( Site 0062), Cheongju-si, North Chungcheong
  - Severance Hospital Yonsei University Health System ( Site 0063), Seoul
- Spain (12):
  - ICO L Hospitalet ( Site 0234), L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario A Coruna ( Site 0239), A Coruña, La Coruna
  - Hospital Universitario Insular de Gran Canaria ( Site 0244), Las Palmas de Gran Canaria, Las Palmas
  - Hospital General Universitario de Valencia ( Site 0231), Valencia, Valenciana, Comunitat
  - Hospital Universitario La Fe ( Site 0233), Valencia, Valenciana, Comunitat
  - Hospital General Universitario de Alicante ( Site 0240), Alicante
  - Hospital Santa Creu i Sant Pau ( Site 0241), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0237), Madrid
  - Hospital Clinico San Carlos ( Site 0235), Madrid
  - Hospital Universitario La Paz ( Site 0236), Madrid
  - Complejo Hospitalario de Malaga ( Site 0238), Málaga
  - Hospital Universitario Miguel Servet ( Site 0242), Zaragoza
- Turkey (Türkiye) (8):
  - Cukurova Universitesi Tıp Fakultesi Balcalı Hastanesi ( Site 0314), Adana
  - Hacettepe Universitesi Tıp Fakultesi ( Site 0316), Ankara
  - Ankara Universitesi Tip Fakultesi. ( Site 0317), Ankara
  - Ankara Sehir Hastanesi ( Site 0323), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0312), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0310), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 0313), Izmir
  - Inonu Universitesi Medical Fakultesi ( Site 0318), Malatya
- United Kingdom (10):
  - Cambridge University Hospitals NHS Trust ( Site 0293), Cambridge, Cambridgeshire
  - North Middlesex University Hospital NHS Trust ( Site 0291), London, London, City of
  - Guys and St Thomas NHS Foundation Trust ( Site 0280), London, London, City of
  - St Georges University Hospitals NHS Foundation Trust. ( Site 0292), London, London, City of
  - Aberdeen Royal Infirmary ( Site 0288), Aberdeen, Scotland
  - Leeds Teaching Hospital NHS Trust. St. James University Hospital ( Site 0276), Leeds
  - Leicester Royal Infirmary ( Site 0284), Leicester
  - Christie NHS Foundation Trust ( Site 0275), Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust ( Site 0286), Metropolitan Borough of Wirral
  - Nottingham City Hospital Campus ( Site 0287), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Herbst RS, Cho BC, Zhou C, Burotto M, Dols MC, Sendur MAN, Moiseyenko V, Casarini I, Nishio M, Hui R, Pons-Tostivint E, Dudnik J, Ahmed S, Okpara CE, Dutcus C, Yin L, Luo Y, Chirovsky D, Bhagwati N, Abreu DR. Lenvatinib Plus Pembrolizumab, Pemetrexed, and a Platinum as First-Line Therapy for Metastatic Nonsquamous NSCLC: Phase 3 LEAP-006 Study. J Thorac Oncol. 2025 Sep;20(9):1302-1314. doi: 10.1016/j.jtho.2025.05.016. Epub 2025 May 24. PMID 40419140
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26810&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with treatment-naïve, metastatic nonsquamous Non-small cell lung cancer (NSCLC) were recruited in this study.
Pre-assignment Details: Per protocol, Part 1 participants were excluded from all Part 2 efficacy and safety outcome measures. China participants randomized during the global study phase (134 participants) were included in all global study analyses. China participants randomized during the China extension phase were excluded from all global study analyses and were included in the China-specific analyses in the extension study (NCT04716933).
Groups:
- Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib: Participants received carboplatin AUC5 or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab 200 mg via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS lenvatinib 8 mg via oral capsule once daily.
- Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib: Participants received carboplatin Area Under Curve 5 mg/mL/min (AUC5) or cisplatin 75 mg/m^2 via intravenous (IV) infusion on Day 1 of each 3-week cycle (Q3W) for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab 200 mg via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS lenvatinib 8 mg via oral capsule once daily.
- Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo: Participants received carboplatin AUC5 or cisplatin 75 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pemetrexed 500 mg/m^2 via IV infusion Q3W for 4 cycles PLUS pembrolizumab 200 mg via IV infusion Q3W for up to 35 cycles (up to 2 years) PLUS placebo matching lenvatinib via oral capsule once daily.
Period: Overall Study
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Started | 13 | 375 | 373
Treated During First Course | 13 | 373 | 372
Treated During Second Course | 1 | 3 | 5
Completed | 0 | 0 | 0
Not Completed | 13 | 375 | 373
Not completed — Sponsor's Decision | 4 | 90 | 102
Not completed — Withdrawal by Subject | 1 | 5 | 4
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 8 | 277 | 266

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo | Total
Number analyzed (Participants) | 13 | 375 | 373 | 761
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (7.6) | 62.0 (9.9) | 63.0 (9.7) | 62.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 121 | 126 | 253
  Male | 7 | 254 | 247 | 508
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 75 | 77 | 152
  Not Hispanic or Latino | 13 | 291 | 279 | 583
  Unknown or Not Reported | 0 | 9 | 17 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 5 | 116 | 114 | 235
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 3
  Black or African American | 0 | 0 | 3 | 3
  White | 8 | 248 | 237 | 493
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 9 | 17 | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by an ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature)
  Participants
    ECOG = 0 | 8 | 135 | 133 | 276
    ECOG = 1 | 5 | 240 | 240 | 485
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Randomization of participants in the study was stratified by PD-L1 tumor proportion score (TPS) at baseline (< 50% or ≥ 50%). Higher percentages of PD-L1 TPS staining correspond to higher positivity of PD-L1 on a tumor.
  Participants
    TPS = < 50% | 10 | 272 | 269 | 551
    TPS = ≥ 50% | 3 | 90 | 91 | 184
    Not Evaluable | 0 | 13 | 13 | 26
Geographic Region [Count of Participants; unit: Participants] — Randomization of participants in this study was stratified by geographic region of the enrolling site (East Asia or non-East Asia).
  Participants
    East Asia | 3 | 111 | 112 | 226
    Non-East Asia | 10 | 264 | 261 | 535

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: Dose-limiting toxicity using Common Terminology Criteria for Adverse Events v4.0 for grading, is defined as any of the following hematologic toxicities: 1) Grade 4 neutropenia, 2) Grade 3 or 4 febrile neutropenia, 3) thrombocytopenia <25,000 cells/mm^3 associated with bleeding and/or which requires platelet transfusion, or any of the following non-hematologic toxicities: 4) any other Grade 4 or 5 toxicity, 5) Grade 3 toxicities lasting >3 days (exclusions apply), 6) Grade 3 hypertension not controlled by medication, 7) Grade 3 or above gastrointestinal perforation, 8) Grade 3 or above wound dehiscence requiring medical or surgical intervention, 9) any grade thromboembolic event, or 10) any Grade 3 nonhematologic laboratory value if medical intervention is required or the abnormality leads to hospitalization.
Time Frame: Cycle 1; each cycle is 21 days (up to 21 days)
Population: The analysis population consisted of all participants enrolled in Part 1 who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib
Number analyzed (Participants) | 13
Participants | 2

2. Primary Outcome: Part 1: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one of more adverse events during Part 1 of this study will be presented.
Time Frame: Up to approximately 48 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib
Number analyzed (Participants) | 13
Participants | 13

3. Primary Outcome: Part 1: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study medication due to and adverse event during Part 1 of this study will be presented.
Time Frame: Up to approximately 58 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib
Number analyzed (Participants) | 13
Participants | 9

4. Primary Outcome: Part 2: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from date of randomization to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. Data are from the product-limit (Kaplan-Meier) method for censored data. PFS as assessed by blinded independent central review (BICR) per RECIST 1.1 is presented.
Time Frame: Up to approximately 36 months
Population: The analysis population consisted of all randomized participants in Part 2 who received at least 1 dose of study intervention and were evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 375 | 373
Months | 12.1 [10.4 to 14.1] | 9.5 [8.3 to 10.7]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and Baseline PD-L1 Status (<50% versus >=50%); Test type: Other; p = 0.07976, Stratified Log Rank; Two-sided p-value based on log-rank test stratified by ECOG performance status, geographic region of the enrolling site, and baseline PD-L1 status; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.74 to 1.05]

5. Primary Outcome: Part 2: Overall Survival (OS)
Description: OS is defined as the time from randomization to the time of death from any cause. OS is presented.
Time Frame: Up to approximately 47 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 375 | 373
Months | 21.8 [18.6 to 24.0] | 22.1 [19.7 to 24.2]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.70818, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.88 to 1.26]

6. Secondary Outcome: Part 2: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. ORR as assessed per modified RECIST 1.1 will be presented.
Time Frame: Up to approximately 19 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 212 | 211
Percentage of Participants | 57.1 [50.1 to 63.8] | 50.7 [43.8 to 57.6]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; Comparison based on Miettinen & Nurminen method stratified by ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and Baseline PD-L1 Status (<50% versus >=50% ); Test type: Other; p = 0.08643, Stratified Miettinen & Nurminen; One-sided p-value for testing. H0: difference in percent = 0 versus H1: difference in percent > 0; Percent Difference = 6.3, 95% CI 2-sided [-2.8 to 15.4]

7. Secondary Outcome: Part 2: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: For participants who demonstrated CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions), DOR is defined as the time from the first documented evidence of CR or PR until PD or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, or death from any cause, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. DOR as assessed per modified RECIST 1.1 will be presented.
Time Frame: Up to approximately 48 months
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 375 | 373
Months | 1.6 [1.1 to 15.4] | 1.6 [1.2 to 20.7]

8. Secondary Outcome: Part 2: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experienced one of more adverse events during Part 2 of this study were presented.
Time Frame: Up to approximately 58 months
Population: The analysis population consisted of all randomized participants in Part 2 who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 373 | 372
Participants | 372 | 370

9. Secondary Outcome: Part 2: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinued study treatment during Part 2 of this study were presented.
Time Frame: Up to approximately 58 months
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 373 | 372
Participants | 127 | 92

10. Secondary Outcome: Part 2: Change From Baseline in Global Health Status (GHS) (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 [EORTC QLQ-C30] Items 29 and 30) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are each scored on a 7-point scale (1=Very poor to 7=Excellent). The two raw scores were averaged into a combined score, then normalized using linear transformation so each participant's score ranged from 0 to 100 (0=Worst overall health/quality of life and 100=Best overall health/quality of life). The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score is presented
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Items 29 and 30 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 369 | 371
Score on a Scale | 0.65 [-1.55 to 2.84] | 1.66 [-0.53 to 3.85]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; Comparision based on a cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors (baseline ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status ( <50% versus ≥50%)) as covariates; Test type: Other; p = 0.4805, t-test, 2 sided; Difference in Least Square Means = -1.01, 95% CI 2-sided [-3.83 to 1.80]

11. Secondary Outcome: Part 2: Change From Baseline in Cough (EORTC Quality of Life Questionnaire-Lung Cancer Module 13 [QLQ-LC13] Item 31) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in cough (EORTC QLQ-LC13 Item 31) score will be presented. A lower score indicates a better outcome.
Time Frame: Baseline and week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 31 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 368 | 371
Score on a scale | -11.77 [-14.72 to -8.81] | -11.47 [-14.42 to -8.53]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.8747, t-test, 2 sided; Difference in Least Square Means = -0.29, 95% CI 2-sided [-3.95 to 3.36]

12. Secondary Outcome: Part 2: Change From Baseline in Chest Pain (EORTC QLQ-LC13 Item 40) Score
Description: The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented. A lower score indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 40 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 368 | 371
Score on a scale | -4.61 [-7.26 to -1.96] | -3.70 [-6.34 to -1.06]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; Comparision based on a cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors (baseline ECOG performance status (0 versus 1), geographic region of the enrolling site (East Asia versus non-East Asia), and baseline PD-L1 Status (<50% versus ≥50%)) as covariates; Test type: Other; p = 0.5941, t-test, 2 sided; Difference in Least Square Means = -0.91, 95% CI 2-sided [-4.24 to 2.43]

13. Secondary Outcome: Part 2: Change From Baseline in Dyspnea (EORTC QLQ-C30 Item 8) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in dyspnea (EORTC QLQ-C30 Item 8) score will be presented. A lower score indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 8 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 369 | 371
Score on a scale | -2.77 [-6.04 to 0.50] | -0.61 [-3.86 to 2.65]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.3115, t-test, 2 sided; covariate = -2.16, 95% CI 2-sided [-6.36 to 2.03]

14. Secondary Outcome: Part 2: Change From Baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) Score
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) score will be presented. A higher score indicates a better quality of life.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Items 1-5 assessment data available.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 369 | 371
Score on a scale | -4.11 [-6.37 to -1.84] | -3.73 [-5.99 to -1.48]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.8134, t-test, 2 sided; covariate = -0.37, 95% CI 2-sided [-3.47 to 2.72]

15. Secondary Outcome: Part 2: Time to True Deterioration (TTD) Based on Change From Baseline in Global Health Status (GHS)/Quality of Life (QoL) (EORTC QLQ-C30 Items 29 and 30) Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in GHS/QoL (EORTC QLQ-C30 Items 29 and 30) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in GHS/QoL score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and Week 27
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 358 | 357
Months | 15.70 [9.66 to NA] — NA=Upper range time to deterioration was not reached at time of data cut-off due to insufficient number of participants experiencing deterioration. | NA [21.32 to NA] — NA=Median and upper range time to deterioration was not reached at time of data cut-off due to insufficient number of participants experiencing deterioration.
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.2133, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.92 to 1.47]

16. Secondary Outcome: Part 2: TTD Based on Change From Baseline in Cough EORTC QLQ-LC13 (Item 31) Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline cough (EORTC QLQ-LC30 Items 31) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in physical functioning score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline And Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-LC30 Item 31 assessment data available at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 356 | 353
Months | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration. | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration.
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.0377, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.02 to 1.94]

17. Secondary Outcome: Part 2: TTD Based on Change From Baseline in Chest Pain EORTC QLQ-LC13 (Item 40) Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline chest pain (EORTC QLQ-C30 Item 40) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in chest pains core, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC QLQ-LC13 chest pain Item 40 Score assessment data available at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 356 | 353
Months | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration. | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration.
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.4084, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.62 to 1.21]

18. Secondary Outcome: Part 2: TTD Based on Change From Baseline in Dyspnea EORTC QLQ-C30 (Item 8) Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline dyspnea (EORTC QLQ-C30 Item 8) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in dyspnea score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Item 8 assessment data available at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 358 | 357
Months | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration. | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration.
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.7955, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.79 to 1.36]

19. Secondary Outcome: Part 2: TTD Based on Change From Baseline in Physical Functioning EORTC QLQ-C30 (Items 1 Through 5) Score
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline physical functioning (EORTC QLQ-C30 Items 1 through 5) score. Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in physical functioning score, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-C30 Items 1 through 5 assessment data available at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 358 | 357
Months | 16.82 [8.84 to 22.51] | NA [NA to NA] — NA=Median, lower and upper range time to deterioration were not reached at time of data cut-off due to insufficient number of participants experiencing deterioration.

20. Secondary Outcome: Part 2: Time to True Deterioration (TTD) Based on Change From Baseline in the Composite Endpoint of Cough (EORTC QLQ-LC13 Item 31), Chest Pain (EORTC QLQ-LC13 Item 40), or Dyspnea (EORTC QLQ-C30 Item 8)
Description: TTD is defined as the time from Baseline to the first onset of a ≥10-point negative change (decrease) from Baseline in the composite endpoint of cough (QLQ-LC13 item 31), chest pain (QLQ-LC13 item 40), or dyspnea (QLQ-C30 Item 8). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The TTD, as assessed based on a ≥10-point negative change (decrease) from Baseline in the composite endpoint of cough, chest pain or dyspnea, will be presented. A longer TTD indicates a better outcome.
Time Frame: Baseline and Week 27
Population: The analysis population consisted of all randomized participants in Part 2 who received at least one dose of study treatment and have at least one EORTC-QLQ-LC13 Items 31 and 40 and EORTC-QLQ-C30 Item 8 assessment data available.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo
Number analyzed (Participants) | 358 | 358
Months | 8.28 [5.98 to 11.07] | 9.33 [7.03 to 12.91]
Statistical Analysis 1: Comparison: Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib vs Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.7191, Stratified Log Rank; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.84 to 1.28]

ADVERSE EVENTS:
Time Frame: Up to approximately 58 months
Description: All-cause mortality was reported on all randomized participants (first and second course). Serious and non-serious AEs were reported among participants who received at least one dose of study treatment. MedDRA preferred terms 'Neoplasm progression', 'Malignant neoplasm progression' and 'Disease progression' not related to the drug were excluded. AEs occurring during second course treatment were collected and presented separately from those occurring during the initial treatment.
Groups:
- Part 1 Second Course: Pembrolizumab Only From Pembrolizumab+Chemotherapy+Lenvatinib: Qualified participants who completed the first course of pembrolizumab plus chemotherapy plus lenvatinib for up to 35 cycles (up to 2 years), but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q2W for up to ~1 year, without chemotherapy plus lenvatinib.
- Part 2 Second Course: Pembrolizumab+Chemotherapy+Lenvatinib: Qualified participants who completed the first course of pembrolizumab plus chemotherapy plus lenvatinib for up to 35 cycles (up to 2 years), but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q2W for up to ~1 year. Participants previously receiving Lenvatinib could continue receiving lenvatinib at investigator's discretion.
- Part 2 Second Course: Pembrolizumab+Chemotherapy+Placebo: Qualified participants who completed the first course of pembrolizumab plus chemotherapy plus lenvatinib for up to 35 cycles (up to 2 years), but experienced disease progression, initiated a second course of pembrolizumab at the investigator's discretion, at 200 mg IV Q2W for up to ~1 year. Participants previously receiving placebo could continue receiving placebo at investigator's discretion.
Arm/Group | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo | Part 1 Second Course: Pembrolizumab Only From Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 Second Course: Pembrolizumab+Chemotherapy+Lenvatinib | Part 2 Second Course: Pembrolizumab+Chemotherapy+Placebo
All-Cause Mortality (participants affected / at risk) | 9/13 | 278/375 | 266/373 | 0/1 | 3/3 | 3/7
Serious Adverse Events (participants affected / at risk) | 7/13 | 232/373 | 189/372 | 1/1 | 1/3 | 3/7
Other Adverse Events (participants affected / at risk) | 13/13 | 366/373 | 363/372 | 1/1 | 2/3 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=13) | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=373) | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo (N=372) | Part 1 Second Course: Pembrolizumab Only From Pembrolizumab+Chemotherapy+Lenvatinib (N=1) | Part 2 Second Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=3) | Part 2 Second Course: Pembrolizumab+Chemotherapy+Placebo (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 17 (19) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 12 (13) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal haematoma (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coeliac artery stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 7 (9) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic haematoma (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 5 (5) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 28 (37) | 36 (40) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 10 (10) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 6 (7) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 10 (10) | 9 (10) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 14 (14) | 15 (16) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 11 (11) | 8 (8) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudocellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 First Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=13) | Part 2 First Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=373) | Part 2 First Course: Pembrolizumab+Chemotherapy+Placebo (N=372) | Part 1 Second Course: Pembrolizumab Only From Pembrolizumab+Chemotherapy+Lenvatinib (N=1) | Part 2 Second Course: Pembrolizumab+Chemotherapy+Lenvatinib (N=3) | Part 2 Second Course: Pembrolizumab+Chemotherapy+Placebo (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 192 (394) | 220 (419) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 26 (30) | 23 (27) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (6) | 84 (104) | 42 (46) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 9 (10) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 9 (9) | 14 (14) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 2 (3) | 24 (25) | 24 (28) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 5 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 33 (47) | 20 (27) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 30 (33) | 18 (20) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (9) | 120 (169) | 110 (143) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (10) | 127 (245) | 69 (107) | 1 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 10 (10) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 23 (25) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 13 (14) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (2) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 11 (15) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (17) | 148 (264) | 137 (246) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 15 (16) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 47 (64) | 21 (30) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 13 (17) | 7 (10) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 69 (133) | 62 (99) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 108 (167) | 110 (175) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (2) | 21 (23) | 25 (29) | 0 (0) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (15) | 116 (182) | 86 (114) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 3 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 7 (11) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (2) | 15 (24) | 15 (18) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (3) | 47 (62) | 28 (35) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 5 (6) | 9 (13) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 7 (7) | 9 (11) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (4) | 61 (81) | 49 (70) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 57 (98) | 61 (83) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (2) | 32 (32) | 23 (24) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 24 (27) | 18 (21) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 10 (13) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 6 (8) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 23 (27) | 21 (22) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 22 (31) | 15 (21) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (11) | 30 (41) | 29 (35) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 132 (271) | 119 (251) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 55 (108) | 55 (95) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 127 (311) | 108 (240) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 31 (52) | 31 (44) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 20 (31) | 9 (18) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (7) | 66 (122) | 69 (104) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 21 (31) | 22 (28) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 23 (31) | 17 (29) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 38 (51) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 49 (73) | 30 (39) | 0 (0) | 0 (0) | 0 (0)
Lactescent serum (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 47 (94) | 43 (82) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 29 (54) | 18 (31) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (6) | 188 (526) | 154 (436) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (4) | 148 (348) | 98 (203) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 69 (82) | 29 (31) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 20 (30) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 119 (372) | 95 (306) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 130 (218) | 112 (150) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (6) | 11 (14) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 39 (69) | 33 (56) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 20 (28) | 19 (26) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 39 (81) | 28 (51) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 19 (26) | 18 (22) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 39 (59) | 27 (41) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2) | 36 (59) | 29 (42) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 44 (72) | 31 (64) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 54 (72) | 33 (38) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 44 (52) | 42 (47) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 19 (20) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 20 (21) | 16 (19) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 32 (43) | 17 (18) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 39 (50) | 36 (42) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 26 (28) | 19 (22) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 45 (64) | 35 (44) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 3 (5) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 20 (23) | 18 (19) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 6 (7) | 8 (10) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 9 (9) | 9 (12) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (5) | 26 (28) | 32 (43) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 10 (11) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (8) | 55 (114) | 26 (37) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 65 (82) | 50 (60) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 31 (36) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 63 (78) | 66 (68) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 55 (86) | 17 (21) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 20 (23) | 14 (20) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 18 (21) | 21 (30) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 20 (21) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (10) | 22 (22) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 15 (19) | 23 (25) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (14) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 16 (19) | 15 (15) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 14 (14) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 13 (13) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 45 (56) | 48 (68) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (7) | 64 (86) | 57 (64) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 9 (10) | 110 (158) | 44 (46) | 0 (0) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Degenerative aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 13 (18) | 12 (21) | 0 (0) | 1 (1) | 0 (0)
Urinary occult blood positive (Investigations) | 0 (0) | 4 (6) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 11 (11) | 9 (20) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (11) | 8 (9) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.

Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT03829319/Prot_SAP_001.pdf